CLINICAL TRIAL: NCT01304225
Title: Panretinal Photocoagulation for Diabetic Retinopathy With PASCAL Laser - an Anatomic and Functional Evaluation of Different Treatment Strategies
Brief Title: Panretinal Photocoagulation for Diabetic Retinopathy With PASCAL Laser
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Renato Magalhães Passos, Doctor at the Ophthalmology Department of UNIFESP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PASCAL-001
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; photocoagulation; PASCAL laser
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100ms single-shot (Active Comparator): Panretinal photocoagulation utilizing 100ms pulse duration, moderate intensity burns, in a single-shot fashion
  Interventions: Procedure: Panretinal photocoagulation
- 20ms multiple-shot (Experimental): Panretinal photocoagulation utilizing 20ms pulse duration, moderate intensity burns, in a multiple-shot fashion
  Interventions: Procedure: Panretinal photocoagulation
- 20ms multiple-shot, barely visible (Experimental): Panretinal photocoagulation utilizing 20ms pulse duration, barely visible intensity burns, in a multiple-shot fashion
  Interventions: Procedure: Panretinal photocoagulation

INTERVENTIONS:
Procedure: Panretinal photocoagulation — Panretinal photocoagulation utilizing 100ms pulse duration, moderate intensity burns, in a single-shot fashion
  Arms: 100ms single-shot
Procedure: Panretinal photocoagulation — Panretinal photocoagulation utilizing 20ms pulse duration, moderate intensity burns, in a multiple-shot fashion
  Arms: 20ms multiple-shot
Procedure: Panretinal photocoagulation — Panretinal photocoagulation utilizing 20ms pulse duration, barely visible intensity burns, in a multiple-shot fashion
  Arms: 20ms multiple-shot, barely visible

SUMMARY:
This study will investigate the clinical efficacy and safety of the PASCAL laser (PAttern SCAn Laser) for diabetic retinopathy. Patients with proliferative or severe nonproliferative retinopathy will be treated with panretinal photocoagulation utilizing different treatment strategies. The investigators believe that using "lower" laser parameters, the clinical response may be equivalent with less adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* proliferative or severe nonproliferative diabetic retinopathy (type 1 or type 2)
* best corrected visual acuity of 20/50 or better
* capability to read and follow instructions
* capability to sign the consignment term

Exclusion Criteria:

* best corrected visual acuity worse than 20/50
* significant macular edema responsible for visual acuity lower than 20/50
* media opacities (includes vitreous hemorrhage in the visual axis, but not a reabsorbing inferior vitreous hemorrhage)
* previous laser treatment (PRP, focal or macular grid)
* glaucoma (confirmed or suspicious)
* other diseases of the retina and optic nerve
* previous ocular surgery in the last 6 months
* impossibility to obtain good quality images of retinography, angiography or OCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe visual loss after 1 year | 1 year
  Severe visual loss is defined as visual acuity worse or equal to 5/200 in two consecutive visits (DRS/ETDRS primary outcome)

SECONDARY OUTCOMES:
Clinical involution of retinal new vessels | 1 year
  Clinical involution of retinal new vessels will be evaluated with retinography and fluorescein angiography
Nerve fiber layer thickness | 1 year
  Nerve fiber layer thickness will be evaluated with Spectral Domain OCT
Retinal sensitivity | 1 year
  Retinal sensitivity will be evaluated with Humphrey computerized perimetry and FDT (Frequency Doubling Technology)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Modi D, Chiranand P, Akduman L. Efficacy of patterned scan laser in treatment of macular edema and retinal neovascularization. Clin Ophthalmol. 2009;3:465-70. doi: 10.2147/opth.s6486. Epub 2009 Aug 20. PMID 19714265
- [Background] Muqit MM, Gray JC, Marcellino GR, Henson DB, Young LB, Patton N, Charles SJ, Turner GS, Dick AD, Stanga PE. In vivo laser-tissue interactions and healing responses from 20- vs 100-millisecond pulse Pascal photocoagulation burns. Arch Ophthalmol. 2010 Apr;128(4):448-55. doi: 10.1001/archophthalmol.2010.36. PMID 20385940
- [Background] Muqit MM, Marcellino GR, Henson DB, Young LB, Patton N, Charles SJ, Turner GS, Stanga PE. Single-session vs multiple-session pattern scanning laser panretinal photocoagulation in proliferative diabetic retinopathy: The Manchester Pascal Study. Arch Ophthalmol. 2010 May;128(5):525-33. doi: 10.1001/archophthalmol.2010.60. PMID 20457972
- [Background] Nagpal M, Marlecha S, Nagpal K. Comparison of laser photocoagulation for diabetic retinopathy using 532-nm standard laser versus multispot pattern scan laser. Retina. 2010 Mar;30(3):452-8. doi: 10.1097/IAE.0b013e3181c70127. PMID 20216293